CLINICAL TRIAL: NCT06611878
Title: Memory for Music: Effects of Individual Intensive Musical Training Based on Singing in Non-musicians With Alzheimer's Disease
Brief Title: Memory for Music: Individual Intensive Musical Training in Alzheimer's Disease
Acronym: M4M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: Universidad de Ciencias Empresariales y Sociales, Buenos Aires, Argentina (Unknown); University of Vienna (Other); University of Bergen (Other); Universidad Nacional de Entre Rios (Other); Kinn Municipality, Norway (Unknown); Oslo Municipality (Other Government); Norwegian Association for Music Therapy (Unknown); Oslo Dementia Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 106684; 344215 (Other Grant/Funding Number: Research Council of Norway)
Record Dates: First submitted 2024-09-05; First posted 2024-09-25 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
Keywords: music and memory; N400; music-based intervention; music therapy; dementia; cognition; mood
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomised crossover design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and instructors cannot be blinded due to the nature of the intervention. External evaluators will remain blinded after randomization; success of blinding will be verified at the end of each participant's participation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive followed by minimal music training (Experimental): Music training conducted by a trained instructor (music therapist or music educator):
  2 sessions per week for 5 months (intensive); no intervention for 2 months (washout period);
  1 session per month for 5 months (minimal).
  Interventions: Behavioral: Music training - intensive; Behavioral: Music training - minimal; Other: Treatment as Usual (TAU)
- Minimal followed by intensive music training (Experimental): Music training conducted by a trained instructor (music therapist or music educator):
  1. session per month for 5 months (minimal); no intervention for 2 months (washout period);
  2. sessions per week for 5 months (intensive).
  Interventions: Behavioral: Music training - intensive; Behavioral: Music training - minimal; Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Music training - intensive — Music training entails learning novel songs the participant chooses from a list. Songs are similar in complexity and length (number of words, high frequency words, harmony, musical complexity, length of verses and chorus). Offering a variety of songs allows to examine memory performance regardless of the specific song chosen. Sessions last 30 to 40 minutes, conducted based on a manual (1. mood observation; 2. warm-up; 3. teaching the chorus, observed liking of song; 4. singing entire chorus; 5. singing chorus in context, 6. session closure with favourite song; 7. final mood observation; session rating), and are video-recorded. External evaluators audit the sessions video recordings to determine adherence to the manual. Sessions are offered twice a week for 5 months.
Behavioral: Music training - minimal — Music training entails learning novel songs the participant chooses from a list. Songs are similar in complexity and length (number of words, high frequency words, harmony, musical complexity, length of verses and chorus). Offering a variety of songs allows to examine memory performance regardless of the specific song chosen. Sessions last 30 to 40 minutes, conducted based on a manual (1. mood observation; 2. warm-up; 3. teaching the chorus, observed liking of song; 4. singing entire chorus; 5. singing chorus in context, 6. session closure with favourite song; 7. final mood observation; session rating), and are video-recorded. External evaluators audit the sessions video recordings to determine adherence to the manual. Sessions are offered once a month for 5 months.
Other: Treatment as Usual (TAU) — Medications, behavioural interventions and other treatments that participants may receive outside the study during the period of participation.

SUMMARY:
This project, called Memory for Music, focuses on the increasing number of people worldwide living with dementia, especially Alzheimer's disease (AD). AD typically starts with memory problems and eventually affects daily activities. Active music interventions, especially singing, have shown positive effects on mood, behavior, and quality of life for people with dementia, but their impact on cognition is not well understood. The project aims to address this gap by studying the effects of learning new songs on cognitive, behavioral, and brain functioning.

The study will involve home-dwelling adults aged 65 or older with AD from Argentina, Austria, and Norway. Participants will undergo 5 months of intensive musical training (twice a week) and 5 months of minimal training (once a month) in a random order, with a 2-month break in between. The interventions include learning new songs with a personal music teacher. General cognition will be measured using the Alzheimer's Disease Assessment Scale - Cognitive (ADAS-cog), and memory for music will be assessed through various methods, including behavioral tasks and brain responses (EEG). Mood will also be evaluated in each session.

The goal is to include 113 participants to ensure reliable detection of meaningful effects. The study will explore how mood and memory for music contribute to changes in cognitive abilities, and whether these effects vary based on factors such as sex, age, AD stage, or previous musical training and general education. The project emphasizes collaboration between researchers, service providers, and users to ensure the study's relevance and applicability.

DETAILED DESCRIPTION:
The number of people living with dementia is increasing and is high in low, middle, and high-income countries. Alzheimer's disease (AD), the most common type of dementia, manifests itself initially with cognitive impairment in memory domains, and later affects all activities of daily living. Active music interventions, particularly singing, can help to improve mood, behaviour problems, and quality of life. Too little is known about their effects on cognition, although some promising studies exist. The M4M project aims to fill this gap by measuring effects of learning new songs on clinical, behavioural and brain functioning. Specifically, M4M aims to examine changes in general cognitive functioning and memory for music in non-musician adults with AD undergoing intensive individual musical training based on singing novel songs, compared to minimal training.

Home-dwelling adults with AD, 65 years or older, in 3 countries (Argentina, Austria, Norway), will receive 5 months of intensive intervention (2x/week) and 5 months of minimal intervention (1x/month), in random order, with a 2-month break in between. Interventions will entail learning new songs with an individual music teacher. At the end of each intervention period, general cognition will be measured with the Alzheimer's Disease Assessment Scale - Cognitive (ADAS-cog) by a person who is unaware of the intervention received. Memory for music will be tested with observations, behavioural tasks, and brain responses (EEG). Mood will be assessed in each session. The investigators aim to include 113 participants; this will help us to reliably detect clinically meaningful effects. The investigators will also examine how mood and memory for music lead to changes in cognitive abilities, and whether effects depend on sex, age, AD stage, or previous musical training or general education. M4M will be conducted in close collaboration between academic researchers, service providers, and service users to ensure relevance and applicability.

Behavioural assessment will be conducted by the instructors and by external evaluators at specific points of the musical training. Mood will be assessed using a 5-point emoji scale, and Sense of Familiarity with the current song will be estimated using a scale that takes into account verbal and behavioural cues; both measures were developed for the purpose of this study.

EEG measures will be collected while participants listen to both unknown melodies and melodies they have learned during the intervention period, and the investigators wish to assess whether in-key violations in known songs will elicit an N400-like event related potential. If participants develop musical semantic memory through our intervention, the investigators expect them to show this N400-like component to in-key violations in familiarized melodies, i.e., those melodies that are introduced and learned during our intervention, but only after the intervention. If an N400 component is detectable during these in-key violations of a newly learned song, it will indicate memory of the new song even if the participant is unable to adhere to a behavioural task or display an observable sense of familiarity. The in-key violations will be introduced at multiple places throughout each melody, which will consist of at least 32 bars. A total of 10 melodies will be played for each participant, of which half are learned in an intervention period (familiarized/to be familiarized). In each of the melodies the investigators will include at least 8 in-key violations. ERPs in response to these in-key violations will be compared to ERPs in response to unchanged notes in structurally similar places in each melody.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease
* Home-dwelling
* Non-musician

Exclusion Criteria:

* Non-Alzheimer dementia
* Living in care home
* History as a professional musician

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
ADAS-cog | 0, 5, 7, 12 months
  ADAS-cog is a scale developed to assess the level of cognitive dysfunction in individuals with Alzheimer's disease.
  The standard ADAS-cog includes the following 11 subtests, with a total scoring range from 0 (no impairment) to 70 (most severe impairments): word recall (0-10); commands (0-5); naming (0-5); constructional praxis (0-5); ideational praxis (0-5); orientation (0-8); word recognition (0-12); remembering word recognition test instructions (0-5); spoken language ability (0-5); comprehension of spoken language (0-5); word-finding difficulty (0-5). The ADAS-cog score is based on the number of errors made within each subtest.
EEG-ERP N400 in response to music stimuli | 0, 5, 7, 12 months
  Electroencephalography (EEG) is a non-invasive method of measuring brain activity. Electrical potential from the brain is measured through electrodes on a cap fitted on the head of the participant. Event-related potentials (ERPs) in response to music violations (unexpected notes in songs) will be analysed to indicate implicit memory for learned music. Generally, ERPs are measured by averaging the EEG signal over multiple repetitions of the same stimulus response. In this study, ERP analyses will focus on amplitude variation of the N400 component, which is a negative inflection of the EEG signal around 400ms after the onset of a stimulus (here an unexpected note in a song presented via audio recording). It is measured in µV and results in a continuous variable. Because the direction of the N400 is negative, and a stronger response indicates better music memory, lower amplitudes values are interpreted as more favourable outcomes.

SECONDARY OUTCOMES:
Mood | Beginning and end of each training session, i.e. min. 1x/month, max. 10x/month, during months 1-5 and 7-12.
  Self-reported mood at beginning and end of each training session, using a 5-point scale with emojis (icons of faces where 1=sad and 5=happy; higher values mean better outcome).
Sense of Familiarity with current song (Instructor) | During each training session, i.e. min. 1x/month, max. 10x/month, during months 1-5 and 7-12.
  Rated by intervention provider during the training session. Ratings for estimated Sense of Familiarity: 1 - None; 2 - Implicit memory, mere exposure effect; 3 - Weak familiarity; 4 - Familiarity; 5 - Weak recollection; 6 - Recollection. For this study, a score of 4 or above is considered as the threshold to determine familiarity-based recognition.
Sense of Familiarity with current song (External Evaluator) | At the end of selected training sessions (last session of each month and when the instructor's rating changes), during months 1-5 and 7-12.
  Rated by an external evaluator based on video recordings of training sessions. Ratings for estimated Sense of Familiarity: 1 - None; 2 - Implicit memory, mere exposure effect; 3 - Weak familiarity; 4 - Familiarity; 5 - Weak recollection; 6 - Recollection. For this study, a score of 4 or above is considered as the threshold to determine familiarity-based recognition.
Performance (chorus solo) | During selected training sessions (last session of each month and when the instructor's rating changes), during months 1-5 and 7-12.
  Performance (independent recall) of a learned song during solo performance, whether the participant needs full support / intermittent support / support in one syllable/word per line / is fully independent. Rated by an external evaluator based on video recordings of training sessions. Possible range 8-32, where highest is best.
Performance (chorus in context) | During selected training sessions (last session of each month and when the instructor's rating changes), during months 1-5 and 7-12.
  Performance (independent recall) of a learned song during performance in context, whether the participant needs full support / intermittent support / support in one syllable/word per line / is fully independent. Rated by an external evaluator based on video recordings of training sessions. Possible range 2-8, where highest is best.
Adverse events | 5, 7, 12 months
  The investigators will ask participants or relatives at each assessment time point about the occurrence and a description of any serious or non-serious adverse events (AEs). Potentially study-related serious AEs, as well as unblinded frequency counts of any AEs, will be shared and discussed with the Data Monitoring and Safety Committee (DSMC) through the trial statistician.

CONTACTS AND LOCATIONS:
Locations (6):
- Universidad de Ciencias Empresariales y Sociales, Buenos Aires, Argentina
- University of Vienna, Vienna, Austria
- Norway (4):
  - University of Bergen, Bergen, Vestland
  - Haraldsplass Diakonale Sykehus, Bergen, Vestland
  - Kinn municipality, Florø
  - Oslo municipality, Oslo

IPD SHARING:
Plan to Share IPD: Yes
Scripting and statistical analysis of baseline and outcome data will be followed by reporting of outcomes in publications and sharing of de-identified individual participant data and analysis code in a public repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication of results; unlimited.
Access Criteria: Open
URL: https://osf.io/tb956/

REFERENCES:
- [Derived] Lichtensztejn M, Cui AX, Geretsegger M, Lundervold AJ, Koelsch S, Pfabigan DM, Assmus J, Langeland E, Ruiz M, Tabernig C, Skogseth RE, Gold C. Memory for Music (M4M) protocol for an international randomised controlled trial: effects of individual intensive musical training based on singing in non-musicians with Alzheimer's disease. BMJ Open. 2025 Oct 20;15(10):e095136. doi: 10.1136/bmjopen-2024-095136. PMID 41120149
- See also: Project website — https://www.memory4music.net/